CLINICAL TRIAL: NCT02930226
Title: A Phase 1, Single-Center, Partial Double-Blind, Randomized, Controlled (Versus Fresh Frozen Plasma [FFP] in Cohort 3 Only) Clinical Study of the Safety of Ascending Doses of Autologous Freeze Dried Plasma (FDP) in Healthy Volunteers
Brief Title: Ascending Doses of Autologous FDP vs FFP
Acronym: FDP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-14-12; IND 17154 (Other: FDA)
Record Dates: First submitted 2016-10-06; First posted 2016-10-12 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Freeze Dried Plasma in Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 1 unit FDP-CPD (Experimental): Subjects are to have sufficient plasma withdrawn during a single WB collection visit to allow re-infusion with 1 unit of autologous FDP-CPD
  Interventions: Biological: Autologous Freeze Dried Plasma (FDP)
- Reinfusion 1 unit FDP-ACD (Experimental): Subjects are to have sufficient plasma withdrawn during 1 plasmapheresis collection visit to allow re-infusion with 1 unit of autologous FDP-ACD
  Interventions: Biological: Autologous Freeze Dried Plasma (FDP)
- Reinfusion 2 units FDP-CPD (Experimental): Subjects are to have sufficient plasma withdrawn during 2 separate WB collection visits to allow re-infusion with 2 units of autologous FDP-CPD
  Interventions: Biological: Autologous Freeze Dried Plasma (FDP)
- Reinfusion 2 units FDP-ACD (Experimental): Subjects are to have sufficient plasma withdrawn during 1 plasmapheresis collection to allow re-infusion with 2 units of autologous FDP-ACD
  Interventions: Biological: Autologous Freeze Dried Plasma (FDP)
- Reinfusion 3 units FDP, 3 units FFP (1st) (Active Comparator): Subjects plasma withdrawn during 2 or 3 plasmapheresis collections to allow re-infusion with 3 units of autologous FDP-ACD and 3 units of autologous control FFP. Subjects will receive in total 6 units over the course of 2 infusion visits. Subjects are to be randomized to treatment schedule arms that dictate the sequence for infusing FDP-ACD and FFP across the 2 infusion visits
  Interventions: Biological: Autologous Freeze Dried Plasma (FDP); Biological: Fresh Frozen Plasma (FFP)
- Reinfusion 3 units FDP, 3 units FFP (2nd) (Active Comparator): Subjects plasma withdrawn during 2 or 3 plasmapheresis collections to allow re-infusion with 3 units of autologous FDP-ACD and 3 units of autologous control FFP. Subjects will receive in total 6 units over the course of 2 infusion visits. Subjects are to be randomized to treatment schedule arms that dictate the sequence for infusing FDP-ACD and FFP across the 2 infusion visits
  Interventions: Biological: Autologous Freeze Dried Plasma (FDP); Biological: Fresh Frozen Plasma (FFP)

INTERVENTIONS:
Biological: Autologous Freeze Dried Plasma (FDP) — Safety of Ascending Doses of Autologous Freeze Dried Plasma (FDP) in Healthy Volunteers
Biological: Fresh Frozen Plasma (FFP) — Controlled FFP in cohort 3 only
  Arms: Reinfusion 3 units FDP, 3 units FFP (1st); Reinfusion 3 units FDP, 3 units FFP (2nd)

SUMMARY:
Assess the safety of single infusions with RePlas FDP product at increasing fixed doses

DETAILED DESCRIPTION:
This is a single-site, partial double-blind study in healthy volunteers designed to assess the safety of infusing ascending doses of reconstituted autologous freeze dried plasma (FDP) in 3 fixed-dose cohorts. Beginning with Cohort 1, subjects will receive a single infusion of 1 unit (approximately 270 mL) of either FDP manufactured from fresh frozen plasma (FFP) derived from autologous whole blood (WB) collection(s) that use citrate phosphate dextrose (CPD) as the anticoagulant (FDP-CPD) or FDP manufactured from FFP units from autologous plasmapheresis where acid citrate dextrose (ACD) is used as the anticoagulant (FDP-ACD). Recruitment of subjects for Cohort 2 follows the completion of infusions in Cohort 1. Subjects in Cohort 2 will receive a single infusion of 2 units (approximately 540 mL) of either FDP-CPD or FDP-ACD before recruitment for Cohort 3 is initiated. Subjects enrolled in Cohort 3 will receive the highest study dose, a plasma infusion dose of 3 units (approximately 810 mL) of FDP-ACD at one infusion visit and the same dose of autologous FFP at another infusion visit. Cohort 3 subjects will only be infused with FDP and FFP products sourced from autologous plasmapheresis. Randomization of Cohort 3 subjects to a treatment sequence determines whether they will be infused with 3 units of FDP or 3 units of FFP at their first infusion visit followed by infusion with the alternate product at the second infusion visit. A 2-week interval will be maintained between infusion visits in Cohort 3. Crossover of FDP and FFP enables comparison of infusion safety and select coagulation factor recoveries within the same subjects between FDP and FFP at this higher dose.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant/non-breastfeeding females;
* Minimum weight is 140 pounds, maximum weight is 220 pounds;
* Ages 18-55 years;
* Self-reports that he or she feels well and healthy;
* Scores ≥ 35 on the Duke Activity Status Index;
* Able to donate 1 unit of WB based on the AABB donor history questionnaire with modifications indicated. Subjects with history of travel which puts them at risk for Creutzfeldt-Jakob Disease (CJD) or malaria will be eligible to participate;
* Has read the educational materials on donating blood and has had his or her questions answered;
* Able and willing to provide written informed consent;
* Available for the duration of the trial, which is approximately 12 weeks for subjects in Cohort 1 and Cohort 2, Arm 4; approximately 16 weeks for Cohort 2, Arm 3 and Cohort 3 (includes time for collections, product manufacture, and infusions), and able to come to the treatment clinic for scheduled study visits;
* Females of childbearing potential should either be surgically sterile (hysterectomy or tubal ligation), or should use a highly effective, medically accepted contraceptive regimen. Highly effective methods of birth control are defined as those which result in a lower failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence, or vasectomized partner;
* All females must have a negative urine pregnancy test prior to enrollment; and
* Understands the English language.

Exclusion Criteria:

* Known liver, kidney, cardiovascular, neurologic, gastrointestinal, blood, endocrine/metabolic, autoimmune or pulmonary disease, or treated or untreated hypertension;
* Cancer of any kind, under treatment or resolved;
* Known or past coagulopathy conditions;
* Any conditions, medications, etc. on the AABB medical deferral list;
* Past history of asthma (defined as use of a prescribed daily asthma controller medication or required asthma medication in the past 2 weeks);
* Past diagnosis of stroke, deep vein thrombosis, or transient ischemic attack
* Family history of venous or arterial thrombosis before the age of 50 in first-degree relatives (i.e., biological parents, full siblings, or children);
* History of abnormal electrocardiogram (EKG);
* Current smoker (defined as having smoked within the last 6 months);
* Known Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS)-related illness or received a positive test result for HIV infection;
* Positive test for Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) or Human T-cell Lymphotropic Virus (HTLV);
* History or significant treated or untreated mental health issues;
* Female subject who is pregnant, lactating, or with a positive pregnancy test;
* Currently taking an antibiotic or another medication for an infection;
* Treatment or use of aspirin (or other platelet inhibiting agents) within 14 days of study donation and infusion visits;
* Currently using any medications for anticoagulant therapy;
* Previous use of clotting factor concentrate(s);
* Receipt of blood or blood products within the past 12 months;
* In the past week, has had a headache and fever at the same time;
* Known intolerance to any excipients (citrate) in the study drug formulation;
* Systolic blood pressure greater than 140 mmHg;
* Diastolic blood pressure greater than 90 mmHg;
* Temperature greater than 100°F;
* Known hematocrit less than 38% for both male and female donors;
* Positive direct antiglobulin test (DAT);
* Treatment with any investigational agent within 1 month before treatment infusion for this trial;
* Participation in any phase of any other investigational trials while participating in this trial;
* Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for follow-up visits on schedule;
* Other unspecified reasons that, in the opinion of the PI, make the subject unsuitable for enrollment; or
* Institutionalized because of legal or regulatory order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Cancelas, MD, PhD, Principal Investigator — Hoxworth Blood Center
Locations (1):
- Hoxworth Blood Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were recruited at an academic medical center between February 2017 and March 2018. The first participant was enrolled on March 6, 2017 and the last participant was enrolled on April 5, 2018.
Pre-assignment Details: Of 40 screened participants, 30 met inclusion criteria and were enrolled. Six participants were withdrawn prior to receiving study treatment. Twenty four participants were infused with plasma.
Groups:
- 1 Unit, Single Infusion FDP-CPD: Subjects are to have sufficient plasma withdrawn during a single WB collection visit to allow re-infusion with 1 unit of autologous FDP-CPD 270 mL
  Autologous Freeze Dried Plasma (FDP): Safety of Ascending Doses of Autologous Freeze Dried Plasma (FDP) in Healthy Volunteers
- 1 Unit, Single Infusion FDP-ACD: Subjects are to have sufficient plasma withdrawn during 1 plasmapheresis collection visit to allow re-infusion with 1 unit of autologous FDP-ACD 270 mL
  Autologous Freeze Dried Plasma (FDP): Safety of Ascending Doses of Autologous Freeze Dried Plasma (FDP) in Healthy Volunteers
- 2 Units, Single Infusion FDP-CPD: Subjects are to have sufficient plasma withdrawn during 2 separate WB collection visits to allow re-infusion with 2 units of autologous FDP-CPD 540 mL
  Autologous Freeze Dried Plasma (FDP): Safety of Ascending Doses of Autologous Freeze Dried Plasma (FDP) in Healthy Volunteers
- 2 Units, Single Infusion FDP-ACD: Subjects are to have sufficient plasma withdrawn during 1 plasmapheresis collection to allow re-infusion with 2 units of autologous FDP-ACD 540 mL
  Autologous Freeze Dried Plasma (FDP): Safety of Ascending Doses of Autologous Freeze Dried Plasma (FDP) in Healthy Volunteers
- 3 Units Per Crossover Infusion FDP-ACD x FFP; 3 Units Per Crossover Infusion FFP x FDP-ACD: Subjects plasma withdrawn during 2 or 3 plasmapheresis collections to allow re-infusion with 3 units of autologous FDP-ACD and 3 units of autologous control FFP. Subjects will receive in total 6 units over the course of 2 infusion visits. Subjects are to be randomized to treatment schedule arms that dictate the sequence for infusing FDP-ACD and FFP across the 2 infusion visits. 810 mL each infusion
  Autologous Freeze Dried Plasma (FDP): Safety of Ascending Doses of Autologous Freeze Dried Plasma (FDP) in Healthy Volunteers
  Fresh Frozen Plasma (FFP): Controlled FFP in cohort 3 only
Period: Overall Study
Arm/Group | 1 Unit, Single Infusion FDP-CPD | 1 Unit, Single Infusion FDP-ACD | 2 Units, Single Infusion FDP-CPD | 2 Units, Single Infusion FDP-ACD | 3 Units Per Crossover Infusion FDP-ACD x FFP | 3 Units Per Crossover Infusion FFP x FDP-ACD
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Technical Problems: Leak in plasma bag | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Unit, Single Infusion FDP-CPD | 1 Unit, Single Infusion FDP-ACD | 2 Units, Single Infusion FDP-CPD | 2 Units, Single Infusion FDP-ACD | 3 Units Per Crossover Infusion FDP-ACD x FFP | 3 Units Per Crossover Infusion FFP x FDP-ACD | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (7.0) | 34.3 (9.9) | 33.5 (4.8) | 33.8 (17.9) | 35.8 (6.1) | 32.0 (10.7) | 34.03 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 0 | 0 | 1 | 3
  Male | 2 | 4 | 4 | 4 | 4 | 3 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 4 | 4 | 4 | 4 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 4 | 4 | 4 | 4 | 4 | 3 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 4 | 4 | 24
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.0 (4.1) | 27.4 (1.3) | 26.2 (4.8) | 26.3 (4.2) | 28.8 (3.6) | 27.8 (2.3) | 27.25 (3.57)
Height [Mean (Standard Deviation); unit: cm] | 172.7 (7.5) | 185.4 (5.5) | 187.3 (8.4) | 177.8 (3.6) | 180.4 (3.6) | 182.2 (11.8) | 180.97 (7.34)
Weight [Mean (Standard Deviation); unit: Kg] | 80.2 (10.3) | 94.1 (7.1) | 91.6 (15.2) | 83.1 (13.4) | 93.4 (8.3) | 92.2 (8.9) | 89.1 (10.86)
Childbearing Potential [Count of Participants; unit: Participants] — Population: Female participants
  Participants
    number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 1 | 3
    Yes | 1 | 0 | 0 | 0 | 0 | 1 | 2
    No | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rh Factor [Count of Participants; unit: Participants]
  Positive | 2 | 4 | 3 | 2 | 3 | 4 | 18
  Negative | 2 | 0 | 1 | 2 | 1 | 0 | 6
Blood Type [Count of Participants; unit: Participants]
  A | 3 | 2 | 3 | 0 | 2 | 2 | 12
  B | 1 | 0 | 0 | 1 | 0 | 0 | 2
  AB | 0 | 1 | 0 | 1 | 0 | 1 | 3
  O | 0 | 1 | 1 | 2 | 2 | 1 | 7
History of any diseases and/or surgeries [Count of Participants; unit: Participants]
  Yes | 3 | 4 | 4 | 3 | 4 | 4 | 22
  No | 1 | 0 | 0 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety of Single Infusions of FDP at Increasing Fixed Doses in Normal Healthy Subjects by Evaluating Vital Signs and Laboratory Tests
Description: Assess the safety of single infusions of FDP at increasing fixed doses of either 1 unit, 2 units, or 3 units in normal healthy subjects by evaluating vital signs during and after infusion
Time Frame: Follow-up assessments on days 2, 8, 29, and telephone assessments on days 3 and 4
Measure: Count of Participants; unit: Participants
Arm/Group | 1 Unit, Single Infusion FDP-CPD | 1 Unit, Single Infusion FDP-ACD | 2 Units, Single Infusion FDP-CPD | 2 Units, Single Infusion FDP-ACD | 3 Units Per Crossover Infusion FDP-ACD x FFP | 3 Units Per Crossover Infusion FFP x FDP-ACD
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
Participants | 4 | 4 | 4 | 4 | 4 | 4

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Assess the safety and tolerability of a fixed-dose infusion of 3 FDP units in comparison to infusion with the same dose of autologous Fresh Frozen Plasma (FFP) in normal healthy subjects by evaluating vital signs and laboratory tests
Time Frame: Follow-up assessments on days 2, 8, 16, 22, 43, and telephone assessments on days 3, 4, 17, and 18
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Units Per Crossover Infusion FDP-ACD x FFP | 3 Units Per Crossover Infusion FFP x FDP-ACD
Number analyzed (Participants) | 4 | 4
Participants | 3 | 1

3. Secondary Outcome: Number of Participants With Significant Changes in Specific Coagulation Values
Description: Determine if the changes in specific coagulation values are similar with clinically meaningful levels pre and post infusion in the different arm groups by evaluating laboratory tests. Blood thrombin, Coombs direct test, Fibrin D dimer, and Thrombin-antithrombin III levels are determined through a blood test to check if your blood is clotting normally. Positive tests or any values below or above the normal reference range is considered abnormal.
Time Frame: For cohorts 1 and 2, follow-up assessments on days 2, 8 and 29. For cohort 3, follow-up assessments on days 2, 8, 16, 22, and 43.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 Unit, Single Infusion FDP-CPD | 1 Unit, Single Infusion FDP-ACD | 2 Units, Single Infusion FDP-CPD | 2 Units, Single Infusion FDP-ACD | 3 Units Per Crossover Infusion FDP-ACD x FFP | 3 Units Per Crossover Infusion FFP x FDP-ACD
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
Participants
  Blood thrombin increased | 0 | 0 | 0 | 0 | 1 | 0
  Coombs direct test positive | 1 | 0 | 0 | 0 | 0 | 0
  Fibrin D dimer increased | 0 | 0 | 0 | 0 | 0 | 1
  Thrombin-antithrombin III increased | 0 | 0 | 0 | 0 | 1 | 0

4. Secondary Outcome: Number of Participants With Significant Changes in Specific Hematology Values
Description: Determine if the changes in specific hematology values are similar with clinically meaningful levels pre and post infusion in the different arm groups by evaluating laboratory tests. The specific hematology values are determined through a blood test. Any values below or above the normal reference range is considered abnormal.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 1 Unit, Single Infusion FDP-CPD | 1 Unit, Single Infusion FDP-ACD | 2 Units, Single Infusion FDP-CPD | 2 Units, Single Infusion FDP-ACD | 3 Units Per Crossover Infusion FDP-ACD x FFP | 3 Units Per Crossover Infusion FFP x FDP-ACD
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Significant Changes in Specific Chemistry Values
Description: Determine if the changes in specific chemistry values are similar with clinically meaningful levels pre and post infusion in the different arm groups by evaluating laboratory tests. Glucose levels and liver function levels, ALT and AST, are determined through a blood test. Any values below or above the normal reference range is considered abnormal.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 1 Unit, Single Infusion FDP-CPD | 1 Unit, Single Infusion FDP-ACD | 2 Units, Single Infusion FDP-CPD | 2 Units, Single Infusion FDP-ACD | 3 Units Per Crossover Infusion FDP-ACD x FFP | 3 Units Per Crossover Infusion FFP x FDP-ACD
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
Participants
  ALT increased | 0 | 1 | 0 | 0 | 0 | 0
  AST increased | 0 | 1 | 0 | 0 | 0 | 0
  Glucose increased | 0 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 11.1 to 25.4 weeks
Arm/Group | 1 Unit, Single Infusion FDP-CPD | 1 Unit, Single Infusion FDP-ACD | 2 Units, Single Infusion FDP-CPD | 2 Units, Single Infusion FDP-ACD | 3 Units Per Crossover Infusion FDP-ACD x FFP | 3 Units Per Crossover Infusion FFP x FDP-ACD
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 2/4 | 0/4 | 0/4 | 4/4 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Unit, Single Infusion FDP-CPD (N=4) | 1 Unit, Single Infusion FDP-ACD (N=4) | 2 Units, Single Infusion FDP-CPD (N=4) | 2 Units, Single Infusion FDP-ACD (N=4) | 3 Units Per Crossover Infusion FDP-ACD x FFP (N=4) | 3 Units Per Crossover Infusion FFP x FDP-ACD (N=4)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Temperature regulation disorder (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Coombs direct test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Blood thrombin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Thrombin-antithrombin III complex increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT02930226/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT02930226/SAP_001.pdf